CLINICAL TRIAL: NCT00117715
Title: Developmental Regulation of CYPs 1A2, 2D6, 3A4
Brief Title: Developmental Regulation of Proteins Responsible for Transforming Drugs in the Body
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Steve Leeder, Pharm.D; Ph.D., Children's Mercy Hospital Kansas City
Other Study IDs: PPRU 10390; Internal IRB #P00 06-46
Record Dates: First submitted 2005-07-06; First posted 2005-07-08 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Developmental regulation of CYPs 1A2, 2D6, 3A4; Ontogeny; pharmacokinetics; drug biotransformation; enzymatic biotransformation of drugs
MeSH Terms: interventions — Genotype; Caffeine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine DNA (source: blood or saliva)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Genotyping and Phenotyping using dextromethorphan and caffeine as probes — Single doses of dextromethorphan (0.3 mg/kg)and caffeine (3.0 mg/kg) are administered and urine is collected overnight for measurement of drug and metabolites to determine drug biotransformation activity.

SUMMARY:
This is a drug metabolism study in one-year old children involving caffeine and dextromethorphan.

DETAILED DESCRIPTION:
For many years, it has been considered dogma that drug biotransformation capability is limited at best in the fetus and newborn but increases over the first year of life to levels in toddlers and young children that generally exceed adult capacity. There are several situations where examination of clinical PK data has revealed discernable patterns of drug clearance that can be attributed to developmental differences in drug biotransformation. It has become apparent that there are developmental differences in expression among drug metabolizing enzyme families (cytochromes P450 or "CYPs", etc.) Furthermore, individual drug metabolizing enzymes with in a family may have unique developmental profiles that influence the therapeutic response, desired or undesired, to a given agent.

All subjects will have a single 5 ml venous blood sample taken upon admission to the study. All subjects will be given a single oral dose of caffeine and dextromethorphan. Patients will be allowed to consume their normal age appropriate diet around the time of study drug administration and through the sample collection periods. All spontaneously voided urine will be collected for a period of 12 hours following the caffeine and dextromethorphan administration

The specific aim of this proposal is to extend the current longitudinal investigation into the preschool age group (1 to 5 years of age). The developmental profile of CYPs, 1A2, 2D6, and 3A4 will be determined by caffeine and dextromethorphan phenotyping procedures. The purpose of this study is to determine the age/developmental stage at which the CYP2 1A2, 2D6 and 3A4 activities exceed adult activities.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 12 months of age at enrollment

Exclusion Criteria:

* Height and weight ratio outside of the 5th to 100th percentile for adjusted age
* Historical and/or biochemical evidence of hepatic, renal, or hematopoetic dysfunction
* Historical or physical evidence of a neurologic disease/condition (excluding simple, febrile seizures)
* Historical or physical evidence of any disorder associated with swallowing and/or gastrointestinal function
* Concomitant therapy with drugs or other products known to alter the activity of hepatic or intestinal microsomal enzymes(e.g., inducers or inhibitors of CYPs 1A2, 2D6, and/or 3A4), P-glycoprotein or potential competing substrates for the CYPs, under study within 7 days of a scheduled phenotyping evaluation
* Evidence of behavioral, developmental, or psychosocial conditions in the subjects and/or parents/caregivers that, in the opinion of the investigator, would have the potential to adversely impact the level of compliance required for successful study completion
* Evidence of geographic instability (i.e., moving of primary residence within last 24 months) that would adversely influence compliance with repeated study visits necessary for completion of the protocol
* Lack of telephone access required to insure adequate subject contact/follow-up
* Inability to obtain written informed consent from the subject's parents/guardians

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children 12 months of age at study entry. Followed longitudinally until 5 uears of age.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2000-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Steven Leeder, Pharm. D, Ph.D., Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Longitudinal Assessment Cohort: Normal healthy children approximately one year of age followed through five years of age to evaluate the ontogeny of CYP1A2, CYP2D6, CYP3A4.
Period: Overall Study
Arm/Group | Longitudinal Assessment Cohort
Started | 121
1 Year | 88
1.5 Year | 85
2 Year | 76
2.5 Year | 70
3 Year | 61
3.5 Year | 60
4 Year | 58
4.5 Year | 55
5 Year | 49
Completed | 49
Not Completed | 72

BASELINE CHARACTERISTICS:
Arm/Group | Longitudinal Assessment Cohort
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.21 (0.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 107
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 58
  White | 46
  More than one race | 6
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in CYP2D6 Drug Metabolism Phenotype With Age
Description: Concentrations of dextromethorphan(DM) and it's metabolite dextrorphan (DX) are quantified in urine and used to estimate the activity of cytochromes P450 2D6 using the well established DM/DX ratio. The longitudinal study design allows for changes in drug metabolism activity as a function of age which can be characterized via least squares regression where the slope of age vs. DM/DX ratio is examined for deviations from zero.
Time Frame: every 6 months for 5 years
Population: Participants completing each milestone visit at each 0.5 years of age.
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | Longitudinal Assessment Cohort
Number analyzed (Participants) | 111
unitless ratio
  Log (DM/DX) Milestone 1: number analyzed (Participants) | 88
  Log (DM/DX) Milestone 1 | -1.974 (0.593)
  Log (DM/DX) Milestone 2: number analyzed (Participants) | 85
  Log (DM/DX) Milestone 2 | -2.083 (0.617)
  Log (DM/DX) Milestone 3: number analyzed (Participants) | 76
  Log (DM/DX) Milestone 3 | -2.162 (0.638)
  Log (DM/DX) Milestone 4: number analyzed (Participants) | 70
  Log (DM/DX) Milestone 4 | -2.073 (0.657)
  Log (DM/DX) Milestone 5: number analyzed (Participants) | 61
  Log (DM/DX) Milestone 5 | -2.161 (0.669)
  Log (DM/DX) Milestone 6: number analyzed (Participants) | 60
  Log (DM/DX) Milestone 6 | -2.185 (0.670)
  Log (DM/DX) Milestone 7: number analyzed (Participants) | 58
  Log (DM/DX) Milestone 7 | -2.284 (0.745)
  Log (DM/DX) Milestone 8: number analyzed (Participants) | 55
  Log (DM/DX) Milestone 8 | -2.177 (0.699)
  Log (DM/DX) Milestone 9: number analyzed (Participants) | 49
  Log (DM/DX) Milestone 9 | -2.384 (0.672)
Statistical Analysis 1: Comparison: Longitudinal Assessment Cohort; Univariate analysis (ANOVA) of the change in log(DM/DX) over time; Test type: Other; p = 0.035, ANOVA — Post-hoc analysis performed using Tukey's Honestly Significant Difference test

2. Primary Outcome: Change in CYP3A4 Drug Metabolism Phenotype With Age
Description: Concentrations of dextromethorphan (DM) metabolites 3-hydroxymorphinan (3HM) and dextrorphan (DX) are quantified in urine and used to estimate the activity of cytochrome P450 3A4 using the well established 3HM/DX ratio. The longitudinal study design allows for changes in drug metabolism activity as a function of age which can be characterized via least squares regression where the slope of age vs. 3HM/DX ratio is examined for deviations from zero.
Time Frame: every 6 months for 5 years
Population: Participants completing each milestone visit at each 0.5 years of age.
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | Longitudinal Assessment Cohort
Number analyzed (Participants) | 111
unitless ratio
  Log (3HM/DX) Milestone 1: number analyzed (Participants) | 85
  Log (3HM/DX) Milestone 1 | -0.069 (0.180)
  Log (3HM/DX) Milestone 2: number analyzed (Participants) | 76
  Log (3HM/DX) Milestone 2 | -0.117 (0.194)
  Log (3HM/DX) Milestone 3: number analyzed (Participants) | 71
  Log (3HM/DX) Milestone 3 | -0.142 (0.223)
  Log (3HM/DX) Milestone 4: number analyzed (Participants) | 70
  Log (3HM/DX) Milestone 4 | -0.158 (0.276)
  Log (3HM/DX) Milestone 5: number analyzed (Participants) | 61
  Log (3HM/DX) Milestone 5 | -0.109 (0.201)
  Log (3HM/DX) Milestone 6: number analyzed (Participants) | 60
  Log (3HM/DX) Milestone 6 | -0.136 (0.194)
  Log (3HM/DX) Milestone 7: number analyzed (Participants) | 58
  Log (3HM/DX) Milestone 7 | -0.133 (0.164)
  Log (3HM/DX) Milestone 8: number analyzed (Participants) | 55
  Log (3HM/DX) Milestone 8 | -0.122 (0.202)
  Log (3HM/DX) Milestone 9: number analyzed (Participants) | 49
  Log (3HM/DX) Milestone 9 | -0.169 (0.218)
Statistical Analysis 1: Comparison: Longitudinal Assessment Cohort; Univariate analysis (ANOVA) of the change in log(3HM/DX) over time; Test type: Other; p = 0.194, ANOVA — Post-hoc analysis performed using Tukey's Honestly Significant Difference test

3. Primary Outcome: Change in CYP1A2 Drug Metabolism Phenotype With Age
Description: Concentrations of caffeine metabolites 5-Acetylamino-6-amino-3-methyluracil (AAMU), 1-methylxanthine (1MX), 1-methyluric acid (1MU), and 1,7-dimethyluric acid (17MU) are quantified in urine and used to estimate the activity of cytochrome P450 1A2 using the well established (AAMU+1MX+1MU)/1,7U ratio. The longitudinal study design allows for changes in drug metabolism activity as a function of age which can be characterized via least squares regression where the slope of age vs. (AAMU+1MX+1MU)/1,7U ratio is examined for deviations from zero.
Time Frame: every 6 months for 5 years
Population: Participants completing each milestone visit at each 0.5 years of age.
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | Longitudinal Assessment Cohort
Number analyzed (Participants) | 111
unitless ratio
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 1: number analyzed (Participants) | 76
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 1 | -0.851 (0.185)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 2: number analyzed (Participants) | 76
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 2 | -0.823 (0.170)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 3: number analyzed (Participants) | 71
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 3 | -0.858 (0.204)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 4: number analyzed (Participants) | 67
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 4 | -0.856 (0.150)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 5: number analyzed (Participants) | 62
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 5 | -0.832 (0.168)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 6: number analyzed (Participants) | 59
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 6 | -0.853 (0.169)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 7: number analyzed (Participants) | 58
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 7 | -0.822 (0.142)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 8: number analyzed (Participants) | 55
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 8 | -0.851 (0.170)
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 9: number analyzed (Participants) | 48
  Log ((AAMU+1MX+1MU)/1,7U) Milestone 9 | -0.821 (0.167)
Statistical Analysis 1: Comparison: Longitudinal Assessment Cohort; Univariate analysis (ANOVA) of the change in log ((AAMU+1MX+1MU)/1,7,U) over time; Test type: Other; p = 0.831, ANOVA — Post-hoc analysis performed using Tukey's Honestly Significant Difference test

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Longitudinal Assessment Cohort
All-Cause Mortality (participants affected / at risk) | 0/111
Serious Adverse Events (participants affected / at risk) | 0/111
Other Adverse Events (participants affected / at risk) | 0/111

LIMITATIONS AND CAVEATS:
Not all enrolled participants were available for evaluation at every milestone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No